CLINICAL TRIAL: NCT06116630
Title: StrokeCog-BBB to Study Cognitive Outcomes Following Stroke
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Manchester (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Marion S Buckwalter, Principal Investigator, Stanford University
Other Study IDs: 63979
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke: Patients who have a history of stroke will be in the first group.
  Interventions: Diagnostic Test: DCE-MRI
- Control: Patients who do not have a history of stroke, but have a history of cardiovascular risk factors will be in the second group.
  Interventions: Diagnostic Test: DCE-MRI

INTERVENTIONS:
Diagnostic Test: DCE-MRI — Both groups will undergo DCE-MRIs.

SUMMARY:
The goal of this observational study is to learn about cognitive outcomes in stroke patients. The main question it aims to answer are: 1. Is blood-brain barrier permeability compromised for years after stroke, 2. Is a blood biomarker of imbalanced angiogenesis dysregulated in chronic stroke and 3. Are there biomarkers that separately or together predicts cognitive decline after stroke, and are other MRI, blood, and clinical characteristics that are associated. Participants will undergo cognitive testing and MRIs two years apart. Researchers will compare cognitive outcomes in non-stroke patients who have cardiovascular risk factors to understand the effects of stroke on these outcomes.

DETAILED DESCRIPTION:
Post-stroke dementia is an important and understudied component of the vascular contributions to cognitive impairment and dementia. Having a stroke approximately doubles the risk of incident dementia for at least a decade afterwards, even after accounting for other vascular risk factors of dementia and the initial effects of the stroke lesion on cognition. Also, silent strokes occur in nearly half of all aging individuals and are associated with dementia. It has been established in wildtype mice that stroke triggers chronic neuroinflammation in the stroke scar and connected brain regions, and that this causes delayed-onset cognitive decline. In humans, there is neuroinflammation in the stroke scar in about half of all chronic stroke survivors on autopsy, even decades after stroke, suggesting it may play a role in people as well. However, there are no biomarkers that can currently be used in living humans to detect who is at risk of cognitive decline and dementia after stroke. The hypothesis to be tested is that inflammation-induced angiogenesis in the stroke and connected regions results in immature leaky vessels that cause blood-brain barrier leakage even very late after stroke. The goal is to establish that there is chronic blood-brain barrier dysfunction after stroke and a dysregulated angiogenesis as a potential mechanism. This would be a fundamental change in how post-stroke dementia is conceptualized and would open avenues for novel therapy development. This will also help better understand vascular contributions to cognitive impairment and dementia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years or over
* One or more vascular risk factors (e.g. high blood pressure, diabetes or vascular disease such as angina, a previous heart attack, a heart bypass or peripheral artery disease in the legs)
* Established vascular disease (previous MI, angina, vascular stent in the peripheral bed)
* Sufficiently fluent in written and spoken English
* Living independently in the community
* Willing/able to give consent to study participation.

Exclusion Criteria:

* Current treatment with IL-1 blockade or established immune-suppressant therapy (e.g. IL-1Ra or IL-1 antibodies), or treatment within the last 3 months
* Currently participating in a clinical trial of investigation medicinal product (CTIMP) or device trial.
* No history of any previous ischaemic or haemorrhagic stroke, a mini-stroke or a serious brain injury
* Do not have dementia
* Renovascular Disease
* Major neurological disease (immune mediated, previous brain tumors)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from Stanford University Hospital, which is a major urban center with a diverse patient population.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of leaky blood vessels in the brain and cognitive scores | 4 years
  Patients will undergo MRI imaging and cognitive testing. Amount of leakage in the blood vessels with be quantified. Scores on the cognitive tests will be normalized with Z scores. The amount of leakage and the z scores will be correlated to better understand the relationship between blood brain barrier leakage and cognition.
Correlation of blood biomarkers and cognitive scores | 4 years
  Blood will be drawn and analyzed for biomarkers, and the biomarkers concentration will be correlated with the z scores from their cognitive tests.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Buckwalter, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No